CLINICAL TRIAL: NCT03316079
Title: Efficacity and Safety of Mechanical Insufflation-exsufflation on Intubated and Mechanically Ventilated Patients
Brief Title: Efficacity and Safety of Mechanical Insufflation-exsufflation on ICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Principal Investigator, Roberto Martinez Alejos, RPT, University Hospital, Bordeaux
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DC2015/02
Record Dates: First submitted 2017-10-03; First posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Mucus Retention; Mechanical Ventilation Complication; Mucus; Plug, Tracheobronchial
Keywords: intensive care; invasive mechanical ventilation; mechanical insufflation-exsufflation; airway mucus clearance; chest physiotherapy; peak expiratory flow; pulmonary mechanics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chest physiotherapy techniques (Active Comparator): Manual chest physiotherapy techniques applied
  Interventions: Other: Chest physiotherapy techniques
- Chest physiotherapy techniques + Mechanical in-exsufflation (Experimental): Mechanical insufflation-exsufflation in addition to manual chest physiotherapy techniques
  Interventions: Device: Mechanical insufflation-exsufflation

INTERVENTIONS:
Other: Chest physiotherapy techniques — Respiratory manual CPT
  Arms: Chest physiotherapy techniques
Device: Mechanical insufflation-exsufflation — CPT + MI-E (4 series of 5 inspiratory-expiratory cycles at +/- 40 cmH2O, 3 seconds of inspiratory time, 2 seconds of expiratory time and 1 second pause between cycles).
  Arms: Chest physiotherapy techniques + Mechanical in-exsufflation

SUMMARY:
Critically ill and intubated patients on mechanical ventilation (IMV) often present retention of respiratory secretions, increasing the risk of respiratory infections and associated morbidity. Endotracheal suctioning (ETS) is the main strategy to prevent mucus retention, but its effects are limited to the first bronchial bifurcation.

Mechanical in-exsufflation devices (MI-E) are a non-invasive chest physiotherapy (CPT) technique that aims to improve mucus clearance in proximal airways by generating high expiratory flows and simulating cough. Currently there are no studies that have specifically assessed the effects of MI-E in critically ill and intubated patients. Thus, the aims of this study are to evaluate efficacy and safety of MI-E to improve mucus clearance in critically ill and intubated patients.

DETAILED DESCRIPTION:
Controlled randomized, cross-over, single blind trial conducted at University Hospital of Bordeaux (France).

Inclusion criteria: Patients (>18 yo) intubated [internal diameter (ID) 7 to 8], sedated [Richmond Agitation Sedation Scale (RASS) -3 to -5], connected to IMV at least 48 h and expected IMV of at least 24h.

Exclusion criteria: Lung disease or pulmonary parenchyma damage, respiratory inspired fraction of oxygen (FiO2) >60% and/or positive end-expiratory pressure (PEEP) > 10 centimetres of water (cmH2O) and/or hemodynamic instability (mean arterial pressure (MAP) < 65 millimetres of mercury (mmHg) although use of vasopressors] , hemofiltered patients through a central jugular catheter, patients on strict dorsal decubitus by medical prescription, and high respiratory infectious risk.

Design: All patients will receive CPT followed by ETS twice daily. However, patients will randomly receive in one of the sessions an additional treatment of MI-E before ETS. MI-E treatment consists in 4 series of 5 in-expiratory cycles at +/- 40 cmH2O, 3 and 2 sec of inspiratory-expiratory time and 1 sec pause between cycles.

Variables: Mucus clearance will be assessed through wet volume of suctioned sputum through a suction catheter connected to a sterile collector container. Pulmonary mechanics will be measured before, after and 1 h post-intervention through a pneumotachograph (PNT). Peak expiratory flow (PEF) generated by MI-E will be continuously measured through a PNT. Hemodynamic measurements will be recorded before, after and 1 h post-intervention.

ELIGIBILITY:
Inclusion criteria :

* Patients over 18 years old.
* Patents endotracheally intubated (tubes between 7mm and 8mm of internal diameter).
* Invasive mechanical ventilation > 48h
* Invasive mechanical ventilation expected > 24h
* RASS between -3 and -5

Exclusion criteria :

* Lung disease with pulmonary parenchyma injury or diseases where mechanical insufflation-exsufflation use is not recommended (eg: emphysema, pneumothorax, pneumomediastinum, hemoptyses, airway instability, acute barotrauma).
* Hemofiltered patients through a central jugular catheter.
* Respiratory instability (FiO2) >60% and/or (PEEP) > 10cmH2O, and/or hemodynamic instability (MAP) < 65mmHg although use of vasopressors)] instability
* Patients on strict dorsal decubitus by medical prescription.
* High risk infection patients (eg: tuberculosis, H1N1) that cannot be disconnected from IMV.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2015-03-06 (Actual); Primary Completion 2017-12-01 (Estimated); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
Mucus volume retrieved | Immediately after treatment
  respiratory secretions (ml) will be suctioned by a suctioning catheter connected to a sterile collector container

SECONDARY OUTCOMES:
Pulmonary mechanics | Immediately before treatment
  Pulmonary mechanics will be measured with a pulmonary mechanics monitor connected to endotracheal tube. We will obtain positive inspiratory pressure (PIP; cmH20), plateau pressure (Ppl; cmH20), tidal volume (Vt; ml). We will combine PIP, Ppl and Vt to obtain static compliance (Cst) (ml/cmH2O).
Pulmonary mechanics | Immediately before treatment
  Pulmonary mechanics will be measured with a pulmonary mechanics monitor connected to endotracheal tube. We will obtain airway resistance (Raw) (cmH2O/l/s).
Pulmonary mechanics | Immediately before treatment
  Pulmonary mechanics will be measured with a pulmonary mechanics monitor connected to endotracheal tube. We will obtain positive inspiratory pressure (PIP; cmH20), positive expiratory pressure (PEEP; cmH20), and peak inspiratory flow (PIF; l/s). We will combine PIP, PEEP and PIF to obtain respiratory system resistance (Rsr) (cmH2O/l/s).
Pulmonary mechanics | Immediately after treatment
  Pulmonary mechanics will be measured with a pulmonary mechanics monitor connected to endotracheal tube. We will obtain airway resistance (Raw) (cmH2O/l/s).
Pulmonary mechanics | Immediately after treatment
  Pulmonary mechanics will be measured with a pulmonary mechanics monitor connected to endotracheal tube. We will obtain positive inspiratory pressure (PIP; cmH20), plateau pressure (Ppl; cmH20), tidal volume (Vt; ml). We will combine PIP, Ppl and Vt to obtain static compliance (Cst) (ml/cmH2O).
Pulmonary mechanics | Immediately after treatment
  Pulmonary mechanics will be measured with a pulmonary mechanics monitor connected to endotracheal tube. We will obtain positive inspiratory pressure (PIP; cmH20), positive expiratory pressure (PEEP; cmH20), and peak inspiratory flow (PIF; l/s). We will combine PIP, PEEP and PIF to obtain respiratory system resistance (Rsr) (cmH2O/l/s).
Pulmonary mechanics | 1 hour after treatment
  Pulmonary mechanics will be measured with a pulmonary mechanics monitor connected to endotracheal tube. We will obtain airway resistance (Raw) (cmH2O/l/s).
Pulmonary mechanics | 1 hour after treatment
  Pulmonary mechanics will be measured with a pulmonary mechanics monitor connected to endotracheal tube. We will obtain positive inspiratory pressure (PIP; cmH20), plateau pressure (Ppl; cmH20), tidal volume (Vt; ml). We will combine PIP, Ppl and Vt to obtain static compliance (Cst) (ml/cmH2O).
Pulmonary mechanics | 1 hour after treatment
  Pulmonary mechanics will be measured with a pulmonary mechanics monitor connected to endotracheal tube. We will obtain positive inspiratory pressure (PIP; cmH20), positive expiratory pressure (PEEP; cmH20), and peak inspiratory flow (PIF; l/s). We will combine PIP, PEEP and PIF to obtain respiratory system resistance (Rsr) (cmH2O/l/s).
Hemodynamic measurements | Immediately before treatment
  Heart Beat per minute (HB) with continous monitoring
Hemodynamic measurements | Immediately after treatment
  Heart Beat per minute (HB) with continous monitoring
Hemodynamic measurements | 1 hour after treatment
  Heart Beat per minute (HB) with continous monitoring
Hemodynamic measurements | Immediately before treatment
  Blood Pressure in mmHg will be measured with continous monitoring
Hemodynamic measurements | Immediately after treatment
  Blood Pressure in mmHg will be measured with continous monitoring
Hemodynamic measurements | 1 hour after treatment
  Blood Pressure in mmHg will be measured with continous monitoring
Arterial blood gases | Immediately before treatment
  pH (in units) will be obtained from radial artery and blood gases analyzed.
Arterial blood gases | Immediately after treatment
  pH (in units) will be obtained from radial artery and blood gases analyzed.
Arterial blood gases | 1 hour after treatment
  pH (in units) will be obtained from radial artery and blood gases analyzed.
Arterial blood gases | Immediately before treatment
  Partial pressure of oxygen (PO2; mmHg) will be obtained from radial artery and blood gases analyzed.
Arterial blood gases | Immediately after treatment
  Partial pressure of oxygen (PO2; mmHg) will be obtained from radial artery and blood gases analyzed.
Arterial blood gases | 1 hour after treatment
  Partial pressure of oxygen (PO2; mmHg) will be obtained from radial artery and blood gases analyzed.
Arterial blood gases | Immediately before treatment
  Partial pressure of carbon dioxide (PCO2; mmHg) will be obtained from radial artery and blood gases analyzed.
Arterial blood gases | Immediately after treatment
  Partial pressure of carbon dioxide (PCO2; mmHg) will be obtained from radial artery and blood gases analyzed.
Arterial blood gases | 1 hour after treatment
  Partial pressure of carbon dioxide (PCO2; mmHg) will be obtained from radial artery and blood gases analyzed.
Arterial blood gases | Immediately before treatment
  Peripheral oxygen saturation (SPO2; %) will be obtained from radial artery and blood gases analyzed.
Arterial blood gases | Immediately after treatment
  Peripheral oxygen saturation (SPO2; %) will be obtained from radial artery and blood gases analyzed.
Arterial blood gases | 1 hour after treatment
  Peripheral oxygen saturation (SPO2; %) will be obtained from radial artery and blood gases analyzed.
Complications | Through study completion
  We will asess the following adverse events that could happen while we will applying protocol:
  * Mean arterial pressure lower than 15% from baseline
  * Systolic blood pressure higher or lower than 15% from baseline
  * Diastolic blood pressure higher or lower than 15% from baseline
  * Heart rate higher or lower than 20% from baseline
  * Oxygen saturation < 85%

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Martinez Alejos, Msc, Principal Investigator — University Hospital Bordeaux, France
Locations (3):
- France (3):
  - Medical ICU, Bordeaux
  - Vascular ICU., Bordeaux
  - Polyvalent ICU. Centre medico-chirurgicale Magellan 2., Pessac

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Konrad F, Schreiber T, Brecht-Kraus D, Georgieff M. Mucociliary transport in ICU patients. Chest. 1994 Jan;105(1):237-41. doi: 10.1378/chest.105.1.237. PMID 8275739
- [Result] American Association for Respiratory Care. AARC Clinical Practice Guidelines. Endotracheal suctioning of mechanically ventilated patients with artificial airways 2010. Respir Care. 2010 Jun;55(6):758-64. PMID 20507660
- [Result] Gosselink R, Bott J, Johnson M, Dean E, Nava S, Norrenberg M, Schonhofer B, Stiller K, van de Leur H, Vincent JL. Physiotherapy for adult patients with critical illness: recommendations of the European Respiratory Society and European Society of Intensive Care Medicine Task Force on Physiotherapy for Critically Ill Patients. Intensive Care Med. 2008 Jul;34(7):1188-99. doi: 10.1007/s00134-008-1026-7. Epub 2008 Feb 19. PMID 18283429
- [Result] Guerin C, Bourdin G, Leray V, Delannoy B, Bayle F, Germain M, Richard JC. Performance of the coughassist insufflation-exsufflation device in the presence of an endotracheal tube or tracheostomy tube: a bench study. Respir Care. 2011 Aug;56(8):1108-14. doi: 10.4187/respcare.01121. PMID 21801577
- [Result] Gomez-Merino E, Sancho J, Marin J, Servera E, Blasco ML, Belda FJ, Castro C, Bach JR. Mechanical insufflation-exsufflation: pressure, volume, and flow relationships and the adequacy of the manufacturer's guidelines. Am J Phys Med Rehabil. 2002 Aug;81(8):579-83. doi: 10.1097/00002060-200208000-00004. PMID 12172066
- [Derived] Martinez-Alejos R, Marti JD, Li Bassi G, Gonzalez-Anton D, Pilar-Diaz X, Reginault T, Wibart P, Ntoumenopoulos G, Tronstad O, Gabarrus A, Quinart A, Torres A. Effects of Mechanical Insufflation-Exsufflation on Sputum Volume in Mechanically Ventilated Critically Ill Subjects. Respir Care. 2021 Sep;66(9):1371-1379. doi: 10.4187/respcare.08641. Epub 2021 Jun 8. PMID 34103385